CLINICAL TRIAL: NCT01860378
Title: Retail Pharmacy Vouchers to Promote Tdap Vaccination for Adults Living With Infants
Brief Title: Vouchers to Promote Tdap Vaccination
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Robert Wood Johnson Foundation (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 13-010045
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Whooping Cough
Keywords: Whooping Cough; Pertussis; Tdap vaccination; Randomized placebo controlled factorial trial
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Video: Full price & $5 off (Active Comparator): Participants will not view the pertussis video
  Interventions: Other: Full price; Other: $5 off
- Video: Full price & $5 off (Experimental): Participants will watch a brief (~ 1 minute) video about Tdap vaccination
  Interventions: Other: Full price; Other: $5 off

INTERVENTIONS:
Other: Full price — Participants will receive a voucher for the full price of a Tdap vaccine ($63.99) + a baby care product voucher or gift card
Other: $5 off — Participants will receive a voucher for $5 off a Tdap vaccine + a baby care product voucher or gift card.

SUMMARY:
This study is a small-scale randomized, placebo-controlled factorial trial of two interventions to increase Tetanus, diphtheria and acellular pertussis (Tdap) immunization rates among infant caregivers. Specifically, the trial will compare a full cost vs. $5 Tdap voucher with or without an educational video.

DETAILED DESCRIPTION:
The incidence of pertussis, a highly contagious respiratory illness, has more than tripled in the past five years, and is on track this year to be the most severe in over a half century. Pertussis is particularly dangerous, and commonly fatal, for young infants who have not completed the primary vaccination series. To protect infants, pregnant women and adult caregivers should receive Tdap vaccination, but coverage is estimated at only 10% for adult caregivers in close contact with infants.

The objective of this study is to conduct a small-scale randomized controlled trial of an intervention to increase Tdap immunization rates among infant caregivers. The intervention is delivered at the newborn primary care visit and consists of two components: (1) Tdap vaccine vouchers redeemable at neighborhood retail pharmacies and (2) video-based education. The vouchers improve vaccine supply by reducing cost and improving accessibility of the vaccine, while the education component increases demand for the vaccine by making salient the dangers of pertussis and the importance adult vaccination to "cocoon" vulnerable infants. We will evaluate the feasibility and acceptability of each component or both compared to none and assess the impact on the vaccination of parents/caregivers of newborn infants.

Recruitment for this pilot study will take place at a pediatric primary care practice site affiliated with a large children's hospital in Philadelphia, Pennsylvania (PA). The practice schedules approximately 135 newborn visits per month, typically at 2-14 days of life. Participants will redeem Tdap vaccine vouchers at 2 local Rite Aid pharmacies which are the closest Rite Aid locations to the clinic site. The pharmacy accepts all major insurance plans, although most plans (including Medicaid) do not cover Tdap vaccine delivered in pharmacies.

All caregivers ≥ 18 years old who accompany an infant to a newborn visit will be approached by the study coordinator and details of the study will be explained. Caregivers will be asked to participate in the study and if interested, informed consent will be obtained before any study related procedures are performed. Potential subjects will then be screened using the protocol inclusion and exclusion criteria. The research assistant will utilize a data collection form to collect demographic data. After completion of the data collection form, participants will view an educational video if randomized to the education arm. After viewing the educational video, or after completion of data collection form for those who were not randomized to video, participants will receive an envelope containing the Tdap and baby care item voucher or gift card.

Unvaccinated caregivers will receive an envelope containing 2 vouchers or a voucher and a gift card. The vouchers are: one for Tdap vaccination and one for a baby care item. Vouchers will be redeemable only at the two participating nearby Rite Aid pharmacies, will have no monetary value, and cannot be redeemed for any items other than the specified vaccine/baby care product.The gift card can be redeemed at any Rite Aid pharmacy.All envelopes will also contain the Center for Disease Control and Prevention (CDC) Vaccine Information Sheet (V.I.S) for the Tdap vaccine. Participants will be randomized to receive either: (1) a voucher for the full price of a Tdap vaccine ($63.99) + a baby care product voucher/or gift card, or (2) a voucher for $5 off a Tdap vaccine + a baby care product voucher/or gift card. The baby care product voucher / gift card will allow us to assess the proportion of respondents who make a trip to one of the pharmacies following the primary care visit and may also increase the probability that the study participants will visit one of the designated retail pharmacies. The full cost voucher removes any cost barriers related to the Tdap vaccine. The $5 voucher allows us to assess the effect of increased awareness, convenience, and accessibility on vaccine uptake, but without a significant price change. If two unvaccinated caregivers accompany an infant and both choose to enroll in the study, they may receive discordant Tdap voucher amounts; however, both will receive baby care product vouchers / gift cards.

Randomization to each arm will occur through block randomization of study numbers that will take place prior to recruitment. The research assistants will show the video and will therefore not be blinded to educational arm. However, research assistants who enroll participants will be blinded to voucher arm as envelopes will be sealed. Research staff will enter the study number on the data collection form but only the principal investigator and study coordinator will have access to the master file indicating allocation to intervention group.

Voucher redemption is voluntary; data regarding vaccination redemption will be collected by Rite Aid pharmacies. Participants who choose to redeem Tdap vaccine vouchers can do so, at their convenience, at 2 local Rite Aid pharmacies. At the pharmacy, the caregiver must complete a screening form before receiving Tdap. Vouchers are serialized with a barcode which is swiped at the time of redemption Baby care item vouchers will be like a coupon and can be redeemed by a cashier at the pharmacy.

Project staff will perform phone follow-up interviews with participants one month after they were enrolled in the study to ascertain vaccination status and to solicit feedback on the intervention and barriers to vaccination.

Baseline characteristics will be summarized by standard descriptive summaries (e.g. means and standard deviations for continuous variables and percentages for categorical variables). All vouchers will have unique identification (ID) numbers. Variables such as age, gender, insurance status, the relationship of the participant(s) to the infant, vaccination status, and the date and time of the voucher distribution will be summarized. The research coordinator will also record how many caregivers refuse to participate or are not approached for enrollment. The proportion of caregivers screened that meet enrollment criteria and the proportion meeting enrollment criteria that consent to participate will be calculated.

We will measure the proportion of participants enrolled that redeemed a study Tdap voucher. In addition, we will assess the feasibility of voucher distribution, the completeness of redemption data recorded at the pharmacy, and the ability to assess caregiver vaccination status. Vaccination status will be determined by self-report at the time of enrollment and at the time of the follow-up interview. Vaccination rates will also be measured by Tdap voucher redemption. We will measure the redemption rate of the Tdap voucher by treatment arm ($5 voucher vs. full-cost voucher, and video vs. no video), adjusting for sociodemographic characteristics. We will also determine the proportion of baby care product vouchers / gift cards redeemed by treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. All caregivers who report that they have never received Tdap
2. Mothers who did not receive Tdap during their most recent pregnancy or since the birth of the child, even if she received Tdap during a previous pregnancy, as Tdap is now recommended for all pregnant women during each pregnancy.
3. Previous receipt of a tetanus containing vaccine (i.e. Td or TT), regardless of the time interval since receipt of the tetanus-containing vaccine will be also eligible for the study.
4. If a participant is certain they have not received Tdap within the past year but uncertain whether he/she has ever received Tdap, we will offer enrollment and encourage participants to obtain immunization records to confirm their status before voucher redemption. Rite Aid will follow their screening procedures which also includes assessing immunization status. Participants who do not know their Tdap vaccination status will receive the voucher intervention.

Exclusion Criteria:

1. Any adult caregiver who has previously received Tdap
2. For recently-pregnant women: If a mother who received Tdap during her most recent pregnancy (2nd trimester or 3rd trimester) or since the birth of the child. Also, if the mother is unsure of her vaccination status and possibly received the vaccine during this pregnancy or in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Rate of Tdap Vaccination | 5 months
  The primary outcome of interest is the difference in vaccination rates between those who received the vouchers vs. those who did not and between those who received the educational video vs. those who did not. We are also interested in measuring whether the educational video acts as an effect modifier in the association between receipt of the voucher and vaccination rates.

SECONDARY OUTCOMES:
Proportion of all vouchers that are redeemed | 5 months
  We will measure the redemption rate of the Tdap voucher by treatment arm ($5 voucher vs. full-cost voucher, and video vs. no video), adjusting for sociodemographic characteristics. We will also determine the proportion of baby care product vouchers redeemed by treatment arm.

OTHER OUTCOMES:
Feasibility of voucher distribution | 5 months
  We will assess the feasibility and acceptability of voucher distribution by measuring the proportion of potential subjects who consent to join the study and are eligible for participation, time required for enrollment, proportion of participants who withdraw from the study, the completeness of redemption data recorded at the pharmacy, and the ability to assess caregiver vaccination status using self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen A Feemster, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Karabots Primary Care Center - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Klein NP, Bartlett J, Rowhani-Rahbar A, Fireman B, Baxter R. Waning protection after fifth dose of acellular pertussis vaccine in children. N Engl J Med. 2012 Sep 13;367(11):1012-9. doi: 10.1056/NEJMoa1200850. PMID 22970945
- [Background] Cherry JD. Epidemic pertussis in 2012--the resurgence of a vaccine-preventable disease. N Engl J Med. 2012 Aug 30;367(9):785-7. doi: 10.1056/NEJMp1209051. Epub 2012 Aug 15. No abstract available. PMID 22894554
- [Background] Healy CM, Rench MA, Baker CJ. Implementation of cocooning against pertussis in a high-risk population. Clin Infect Dis. 2011 Jan 15;52(2):157-62. doi: 10.1093/cid/ciq001. PMID 21288837
- [Background] Centers for Disease Control and Prevention (CDC). Pertussis--United States, 1997-2000. MMWR Morb Mortal Wkly Rep. 2002 Feb 1;51(4):73-6. PMID 11837909
- [Background] Bisgard KM, Pascual FB, Ehresmann KR, Miller CA, Cianfrini C, Jennings CE, Rebmann CA, Gabel J, Schauer SL, Lett SM. Infant pertussis: who was the source? Pediatr Infect Dis J. 2004 Nov;23(11):985-9. doi: 10.1097/01.inf.0000145263.37198.2b. PMID 15545851
- [Background] Wendelboe AM, Njamkepo E, Bourillon A, Floret DD, Gaudelus J, Gerber M, Grimprel E, Greenberg D, Halperin S, Liese J, Munoz-Rivas F, Teyssou R, Guiso N, Van Rie A; Infant Pertussis Study Group. Transmission of Bordetella pertussis to young infants. Pediatr Infect Dis J. 2007 Apr;26(4):293-9. doi: 10.1097/01.inf.0000258699.64164.6d. PMID 17414390
- [Background] Centers for Disease Control and Prevention (CDC). Updated recommendations for use of tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine (Tdap) in pregnant women and persons who have or anticipate having close contact with an infant aged <12 months --- Advisory Committee on Immunization Practices (ACIP), 2011. MMWR Morb Mortal Wkly Rep. 2011 Oct 21;60(41):1424-6. PMID 22012116
- [Background] Centers for Disease Control and Prevention (CDC). Updated recommendations for use of tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis (Tdap) vaccine in adults aged 65 years and older - Advisory Committee on Immunization Practices (ACIP), 2012. MMWR Morb Mortal Wkly Rep. 2012 Jun 29;61(25):468-70. PMID 22739778
- [Background] Advisory Committee on Immunization Practices. Recommended adult immunization schedule: United States, 2012. Ann Intern Med. 2012 Feb 7;156(3):211-7. doi: 10.7326/0003-4819-156-3-201202070-00388. Epub 2012 Jan 31. No abstract available. PMID 22298576
- [Background] Lessin HR, Edwards KM; Committee On Practice And Ambulatory Medicine; Committee On Infectious Diseases. Immunizing parents and other close family contacts in the pediatric office setting. Pediatrics. 2012 Jan;129(1):e247-53. doi: 10.1542/peds.2011-2937. Epub 2011 Dec 26. PMID 22201157
- [Background] Centers for Disease Control and Prevention (CDC). Adult vaccination coverage--United States, 2010. MMWR Morb Mortal Wkly Rep. 2012 Feb 3;61(4):66-72. PMID 22298302
- [Background] Walter EB, Allred N, Rowe-West B, Chmielewski K, Kretsinger K, Dolor RJ. Cocooning infants: Tdap immunization for new parents in the pediatric office. Acad Pediatr. 2009 Sep-Oct;9(5):344-7. doi: 10.1016/j.acap.2009.05.027. Epub 2009 Jul 12. PMID 19596219
- [Background] Bearden DT, Holt T. Statewide impact of pharmacist-delivered adult influenza vaccinations. Am J Prev Med. 2005 Dec;29(5):450-2. doi: 10.1016/j.amepre.2005.08.003. PMID 16376709
- [Background] Eades CE, Ferguson JS, O'Carroll RE. Public health in community pharmacy: a systematic review of pharmacist and consumer views. BMC Public Health. 2011 Jul 21;11:582. doi: 10.1186/1471-2458-11-582. PMID 21777456
- [Background] Crawford ND, Blaney S, Amesty S, Rivera AV, Turner AK, Ompad DC, Fuller CM. Individual- and neighborhood-level characteristics associated with support of in-pharmacy vaccination among ESAP-registered pharmacies: pharmacists' role in reducing racial/ethnic disparities in influenza vaccinations in New York City. J Urban Health. 2011 Feb;88(1):176-85. doi: 10.1007/s11524-010-9541-6. PMID 21279450